CLINICAL TRIAL: NCT07289347
Title: EFFECT OF A LIGHT STIMULATED FOOTSTEPS PATHWAY ON KINEMATICS OF GAIT IN SPASTIC DIPLEGIC CHILDREN
Brief Title: EFFECT OF A LIGHT STIMULATED FOOTSTEPS PATHWAY ON GAIT IN SPASTIC CHILDREN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amira saad mohamed (Other)
Responsible Party: Sponsor-Investigator, Amira saad mohamed, lecturer of physical therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/006097
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spastic Diplegia
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): This group of fifteen children received a regular traditional therapeutic exercise program based on the Pragmatic approach.
  Interventions: Other: therapeutic exercise
- Group B (Experimental): The fifteen children in this group got the same therapeutic exercise program as the control group, as well as 30 minutes of gait training on light stimulated footsteps pathway.
  Interventions: Other: therapeutic exercise; Other: gait training on light stimulated footsteps pathway

INTERVENTIONS:
Other: therapeutic exercise — Balance training from different positions. Weight shifting exercises by facilitation of single limb support while standing.
  Ascending and descending stairs. Gait training between parallel bars
Other: gait training on light stimulated footsteps pathway — same routine program as the control group as well as 30 minutes of gait training on light stimulated footsteps pathway:
  1. Walk on the light stimulated footsteps (Forward steps)
  2. Walk on the light stimulated footsteps (backward steps)
  3. Tandem gait over light yellow line
  Arms: Group B

SUMMARY:
PURPOSE: The purpose of this study will be investigation of the effect oflight stimulated footsteps pathway on kinematics of gait in spastic diplegic children BACKGROUND: The goal of most therapy procedures for children with spastic cerebral palsy is to increase their walking abilities. Locomotor training usinglight stimulated footsteps pathwayhas been recommended for the rehabilitation of children with cerebral palsy in an effort to improve walking independence and gait speed.

HYPOTHESES: Walking on light stimulated footsteps pathway may not affect kinematics of gait in spastic diplegic children RESEARCH QUESTION: Does walking on light stimulated footsteps pathway have any effect onkinematics of gait in spastic diplegic children?

ELIGIBILITY:
Inclusion Criteria:

* Age will range between5 and 8 years old.
* They had Grade 1 and 1+ hypertonia according to Modified Ashworth Scale (Bohannon and Smith, 1987)
* Motor Classification System, they were at level I and II (GMFCS)
* They will capable of following commands and comprehend them.
* They will exhibit defective gait kinematics, which can be determined through gait kinematics evaluation.
* All patients who will be enrolled to the study will have their informed consent.

Exclusion Criteria:

* Epilepsy history.
* Taking any anti spastic drugs.
* Both lower limbs had permanent deformity.
* Surgical intervention history.
* Have visual or auditory defects.
* Chest infections or unstable cardiac status.
* Infective skin conditions.
* Markedly high or low blood pressure.
* Individuals with cardiopulmonary conditions.
* Individuals with any pelvic disease.
* Individuals undergoing radiation therapy or chemotherapy.
* Hepatic or pancreatic diseases.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-09-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
step length | At baseline and re assessed following 3 months
  kinovea software used to evaluate step length The unit of measurement for Step Length is centimeter (cm)
step width | At baseline and re assessed following 3 months
  kinovea software used to evaluate step width The unit of measurement for Step width is centimeter (cm)
spasticity | At baseline and re assessed following 3 months
  The Modified Ashworth Scale (MAS) used for evaluation
  MAS assigns a grade of spasticity from a 0-4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch.
gross motor function | At baseline and re assessed following 3 months
  The Gross Motor Function Measure (GMFM) is a standardized tool used to assess changes in gross motor function in children, particularly those with cerebral palsy.
  The GMFM uses a four-point ordinal scale for scoring each item, where:
  0: Does not initiate
  1. Initiates (but does not complete)
  2. Partially completes
  3. Completes the task fully Scores can be summed to calculate raw and percent scores for each dimension and a total GMFM score.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt